CLINICAL TRIAL: NCT05128864
Title: Prospective, Randomized, Double Blinded Trial Comparing Clinical, Radiological and Laboratory Outcomes of Hight Tibial Osteotomy With or Without Concomitant Fulkerson Osteotomy
Brief Title: High Tibial Osteotomy With/Without Fulkerson Osteotomy in Knee OA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Rafał Kamiński, Chair of Division, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: HTO_fulkerson
Record Dates: First submitted 2020-07-18; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis, Knee; Patellofemoral Disorder
Keywords: HTO; Fulkerson; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HTO and Fulkerson (Active Comparator): High Tibial Osteotomy with Antero-medialisation of Tibial Tubercle
  Interventions: Procedure: High Tibial Osteotomy
- HTO (Sham Comparator): Descending Hight Tibial Osteotomy
  Interventions: Procedure: High Tibial Osteotomy

INTERVENTIONS:
Procedure: High Tibial Osteotomy — Surgery procedure - High Tibial Osteotomy

SUMMARY:
This study will compare Hight Tibial Osteotomy with or without Fulkerson Osteotomy performed on patients with early stages of Osteoarthritis with patellofemoral joint disorders. The purpose of this study is evaluate which type of osteotomy provides better clinical, radiological and laboratory outcomes.

DETAILED DESCRIPTION:
Progression of knee cartilage degenerative changes leads to necessary total knee arthroplasty in future, which is the most popular procedure for treating OA. HTO applied at early stages of osteoarthritis allow slow down cartilage degeneration process, but the choice of performed surgery depends on surgeons personal assessment. Patellofemoral Pain Syndrome often occurs with knee arthritis. Antero-medialisation of tibial tubercle is frequent procedures for patella maltracking. So far, both, HTO and Fulkerson osteotomy was performed separately, even if patient have symptoms from patellofemoral joint and OA. The investigators believe that simultaneously surgery of HTO and fulkerson Osteotomy provides better outcomes and significantly slow down knee degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Knee medial compartment or patellofemoral osteoarthritis in medical interview and physical examination
* Confirmation of cartilage degeneration/damage and knee malalignment in radiological tests

Exclusion Criteria:

* no informed consent to participate in the study
* age under 18 years or above 65
* multi ligament injury or single plane knee instability
* another musculoskeletal disorders in lower limb
* lower limb deformity requiring axis correction below 4o or above 12.5o
* joints inflammatory diseases
* ASA score > II

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Biomechanics MRI | 1 year
  Patellofemoral Joints Biomechanics improvement measured
Biomechanics MRI | 2 years
  Patellofemoral Joints Biomechanics improvement measured
Biomechanics X-ray | 12 weeks
  Patellofemoral Joints Biomechanics improvement measured
Biomechanics X-ray | 6 months
  Patellofemoral Joints Biomechanics improvement measured
Biomechanics X-ray | 12 months
  Patellofemoral Joints Biomechanics improvement measured
Biomechanics X-ray | 24 months
  Patellofemoral Joints Biomechanics improvement measured

SECONDARY OUTCOMES:
KOOS | 12 weeks
  Knee Injury and Osteoarthritis Outcome Score
KOOS | 6 months
  Knee Injury and Osteoarthritis Outcome Score
KOOS | 12 months
  Knee Injury and Osteoarthritis Outcome Score
KOOS | 24 months
  Knee Injury and Osteoarthritis Outcome Score
IKDC | 12 weeks
  International Knee Documentation Committee
IKDC | 6 months
  International Knee Documentation Committee
IKDC | 12 months,
  International Knee Documentation Committee
IKDC | 24 months
  International Knee Documentation Committee
Tegner Lysholm | 12 weeks,
  Tegner Lysholm Knee Scoring Scale
Tegner Lysholm | 6 months
  Tegner Lysholm Knee Scoring Scale
Tegner Lysholm | 12 months
  Tegner Lysholm Knee Scoring Scale
Tegner Lysholm | 24 months
  Tegner Lysholm Knee Scoring Scale
SF-36 | 12 weeks
  The Short Form (36) Health Survey
SF-36 | 6 months
  The Short Form (36) Health Survey
SF-36 | 12 months
  The Short Form (36) Health Survey
SF-36 | 24 months
  The Short Form (36) Health Survey
VAS | 12 week
  Pain Visual Analog Scale
VAS | 6 months
  Pain Visual Analog Scale
VAS | 12 months
  Pain Visual Analog Scale
VAS | 24 months
  Pain Visual Analog Scale
Blood test | 2nd day
  CRP, IL-6, CTx
Blood test | 6 weeks
  CRP, IL-6, CTx

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Kaminski, Principal Investigator — PCME, Otwock, Poland
Locations (1):
- Department of Orthopaedics and Traumatology, Postgraduate Center for Medical Education, Professor A. Gruca Teaching Hospital, Otwock, Masovian Voivodeship, Poland